CLINICAL TRIAL: NCT07327086
Title: Evaluation of Serum Chromium, Nickel, and Magnesium Levels in Patients With Type 2 Diabetes Mellitus and Periodontitis: A Cross-Sectional Study
Brief Title: Serum Chromium, Nickel, and Magnesium in Type 2 Diabetic Periodontitis
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra Bozkurt, Assistant Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: 2025/172
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Periodontal Disease
Keywords: Periodontal disease; Trace Elements; Type 2 Diabetes Mellitus; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontal Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group: Systemically and periodontally healthy individuals.
  Interventions: Other: No intervention (Observational study)
- Periodontitis group: Systemically healthy individuals with Stage II, Grade B periodontitis.
  Interventions: Other: No intervention (Observational study)
- Controlled T2DM with periodontitis group: Individuals with HbA1c < 7.0 and Stage II, Grade B periodontitis.
  Interventions: Other: No intervention (Observational study)
- Uncontrolled T2DM with periodontitis group: Individuals with HbA1c ≥ 7.0 and Stage II, Grade C periodontitis.
  Interventions: Other: No intervention (Observational study)

INTERVENTIONS:
Other: No intervention (Observational study) — Participants were not assigned to any therapeutic or preventive intervention. The study involved periodontal examination and blood sample collection for serum trace element analysis only.

SUMMARY:
Periodontitis is a chronic immunoinflammatory disease that has been increasingly associated with systemic conditions, particularly type 2 diabetes mellitus (T2DM). Trace elements such as chromium (Cr), magnesium (Mg), and nickel (Ni) play important roles in metabolic regulation, insulin signaling, inflammatory responses, and tissue integrity. Alterations in the serum levels of these elements have been reported in T2DM; however, their relationship with periodontal status remains poorly understood. This cross-sectional observational study aims to evaluate serum Cr, Mg, and Ni levels in individuals with T2DM and chronic periodontitis and to investigate their potential associations with periodontal clinical parameters.

DETAILED DESCRIPTION:
Detailed Description

Periodontal diseases are chronic immunoinflammatory conditions initiated by the interaction between the microbial dental plaque biofilm and the host immune response, leading to progressive destruction of the alveolar bone and connective tissues. Although traditionally considered localized oral infections, increasing evidence indicates that periodontitis has significant systemic implications. A well-established bidirectional relationship exists between periodontitis and type 2 diabetes mellitus (T2DM), with periodontitis being recognized as the sixth complication of diabetes. Both conditions are characterized by elevated proinflammatory cytokines and mediators, which may mutually exacerbate disease severity and progression.

Chromium (Cr) is an essential trace element involved in carbohydrate and lipid metabolism and plays a key role in insulin signaling by enhancing insulin receptor activity through its interaction with chromodulin. Chromium deficiency has been proposed as a potential risk factor for the development of diabetes, and chromium supplementation has been reported to improve glycemic control in some individuals with T2DM. Although limited studies suggest alterations in salivary chromium levels in patients with chronic periodontitis, possibly due to periodontal tissue breakdown or metal release from restorative materials, the association between periodontal disease and serum chromium levels has not been directly investigated to date.

Magnesium (Mg) is a vital mineral acting as a cofactor for more than 300 enzymatic reactions and is essential for energy metabolism, oxidative phosphorylation, and membrane integrity. Reduced serum magnesium levels are commonly observed in individuals with T2DM, and magnesium deficiency has been associated with impaired glucose-insulin metabolism and enhanced inflammatory responses. Experimental and clinical studies suggest that magnesium deficiency may aggravate periodontal inflammation and negatively affect periodontal tissue healing; however, studies evaluating magnesium status in individuals with concomitant T2DM and chronic periodontitis are limited.

Nickel (Ni) is a widely distributed environmental heavy metal, and human exposure occurs through air, water, food, tobacco products, dental materials, and metal alloys. Evidence regarding the association between nickel exposure and diabetes is inconsistent, with some studies reporting no association and others suggesting an increased risk of diabetes with higher nickel exposure. To date, no studies have directly evaluated the relationship between periodontal disease and serum nickel levels.

Given the complex interactions among trace elements in metabolic and inflammatory pathways, the simultaneous evaluation of serum chromium, magnesium, and nickel levels may provide valuable insights into the pathophysiology of T2DM and chronic periodontitis. However, current literature lacks studies assessing these three elements together in individuals with T2DM and chronic periodontitis.

This cross-sectional observational study was conducted in accordance with the Declaration of Helsinki and approved by the Kahramanmaraş Sütçü İmam University Medical Faculty Ethics Committee. Adult participants were recruited from individuals undergoing systemic evaluation at the Department of Endocrinology and Metabolism and subsequently referred for periodontal examination. Eligible participants were allocated into four groups based on systemic and periodontal status: periodontally and systemically healthy controls, systemically healthy individuals with chronic periodontitis, individuals with controlled T2DM and chronic periodontitis, and individuals with uncontrolled T2DM and chronic periodontitis.

Comprehensive periodontal examinations were performed by a calibrated examiner using standard clinical indices, including plaque index, gingival index, bleeding on probing, probing pocket depth, and clinical attachment level. Periodontal diagnoses were established according to the 2017 World Workshop Classification of Periodontal and Peri-Implant Diseases and Conditions. Fasting venous blood samples were collected, and serum chromium, magnesium, and nickel levels were analyzed using atomic absorption spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Having at least 20 natural teeth, excluding third molars
* Diagnosed with type 2 diabetes mellitus or systemically healthy, according to group allocation
* Willingness to participate in the study and provision of written informed consent

Exclusion Criteria:

* Presence of systemic diseases other than type 2 diabetes mellitus (e.g., renal or hepatic failure, cardiovascular disease, organ transplantation, or current or previous cancer treatment)
* Use of antibiotics, non-steroidal anti-inflammatory drugs, corticosteroids, immunosuppressive drugs, calcium channel blockers, beta blockers, oral contraceptives, or anticoagulants within the last 3 months
* History of non-surgical periodontal treatment within the last 6 months or periodontal surgery within the last 12 months
* Pregnancy or lactation
* Body mass index (BMI) ≥ 30 kg/m²
* Current smoking or alcohol consumption
* Use of vitamin, mineral, or antioxidant supplements within the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult individuals aged 18 years and older who were systemically evaluated at the Department of Endocrinology and Metabolism and subsequently referred for periodontal examination. Participants include systemically and periodontally healthy individuals as well as patients diagnosed with chronic periodontitis, with or without type 2 diabetes mellitus. Eligible participants were allocated into study groups based on periodontal status and glycemic control.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Serum levels of chromium, magnesium, and nickel | Single time point (cross-sectional assessment)
  The primary outcome is the assessment of fasting serum chromium, magnesium, and nickel concentrations measured using atomic absorption spectrometry in individuals with type 2 diabetes mellitus with and without chronic periodontitis, and systemically healthy controls.

SECONDARY OUTCOMES:
Periodontal clinical parameters | Single time point
  Plaque index, gingival index, bleeding on probing, probing pocket depth, and clinical attachment level assessed during periodontal examination.
Association between serum trace element levels and periodontal parameters | Single time point
  Evaluation of correlations between serum chromium, magnesium, and nickel levels and periodontal clinical measurements.
Effect of glycemic control on serum trace element levels | Single time point
  Comparison of serum chromium, magnesium, and nickel levels between controlled (HbA1c < 7.0) and uncontrolled (HbA1c ≥ 7.0) type 2 diabetes mellitus groups.

CONTACTS AND LOCATIONS:
Overall Officials: esra bozkurt, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers, as there is no predefined data-sharing plan in the study protocol or informed consent, and all data will be used solely for the purposes of the present research in accordance with ethical approval and data protection regulations.

REFERENCES:
- [Result] Titcomb TJ, Liu B, Lehmler HJ, Snetselaar LG, Bao W. Environmental Nickel Exposure and Diabetes in a Nationally Representative Sample of US Adults. Expo Health. 2021 Dec;13(4):697-704. doi: 10.1007/s12403-021-00413-9. Epub 2021 Sep 29. PMID 35685677
- [Result] Toaima DN, Abdel-Maksoud KS, Atef HM, Salah NY. Magnesium, fibrinolysis and clotting interplay among children and adolescents with type 1 diabetes mellitus; potential mediators of diabetic microangiopathy. Nutr Diabetes. 2025 Apr 1;15(1):13. doi: 10.1038/s41387-025-00368-9. PMID 40169565
- See also: Kahramanmaraş Sütçü İmam University Medical Research Ethics Committee — https://tipfakultesi.ksu.edu.tr/Default.aspx?SId=5407